CLINICAL TRIAL: NCT05276206
Title: Comparative Study Between Transversus Abdominus Plain Block, Local Subcutaneous Injection in the Wound, and Intravenous Nalbuphine in Decreasing Postoperative Pain in Cesarean Section
Brief Title: Application of Transversus Abdominus Plain Block, Local Subcutaneous Injection and IV Nalbuphine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Mahmoud Raslan
Record Dates: First submitted 2022-02-20; First posted 2022-03-11 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Post Operative Pain; Cesarean Section Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- NSAID (Active Comparator): The Control group will be given nothing and only non-steroidal anti-inflammatory drugs on need
  Interventions: Drug: NSAID , NALUFIN , local anesthetic andTAP Block
- Nalufin (Active Comparator): group will be given IV nalufin
  Interventions: Drug: NSAID , NALUFIN , local anesthetic andTAP Block
- local anesthetic group (Active Comparator): the local anesthetic group will be given a S.C injection of local anesthetic in the wound
  Interventions: Drug: NSAID , NALUFIN , local anesthetic andTAP Block
- TAP block (Active Comparator): Total abdominal plain block group will be given a TAP block
  Interventions: Drug: NSAID , NALUFIN , local anesthetic andTAP Block

INTERVENTIONS:
Drug: NSAID , NALUFIN , local anesthetic andTAP Block — The pain level of the cases is evaluated by means of the digital pain (numeric rating) scale from 0 to 10 in which 0 means "no pain" and 10 means "the worst pain" as well as the duration of pain relief and the need for another dose of the same analgesic or other. The pain level is evaluated again if it is present.
  In all groups non steroidal anti-inflammatory drugs will be given as a rescue analgesic and the total dose will be calculated and compared

SUMMARY:
Approximately 1 in 5 women who undergo CS will experience severe acute postoperative pain. The severity of pain in the acute postoperative period is a significant predictor for the development of chronic pain, which occurs in 9.2%-18% of women who undergo CS. Furthermore, severe acute post-cesarean pain triples a woman's risk of developing postpartum depression and negatively affects breastfeeding and infant care. For these reasons, it is imperative to provide adequate postoperative analgesia in this patient population

DETAILED DESCRIPTION:
Local wound infiltration is an attractive strategy since it is efficacious and side effects are minimal. Nowadays, there is a trend toward preferring ropivacaine over other local anesthetic agents due to the longer duration of action and better safety profile. Local anesthetic infiltration, however, has a limitation in that pain relief is offered till the effects of local anesthetic action lasts. Efforts are being made to prolong the duration of action of local anesthetic skin infiltration, and dexmedetomidine is one such agent which can potentiate and prolong the duration of local anesthetic wound infiltration for pain relief.

A transversus abdominis plane (TAP) block provides analgesia of the anterior and lateral abdominal wall below the umbilicus by blocking the T6-L1 segmental nerves as they lie within the fascial plane between the transversus abdominis and internal oblique muscles: bilateral block for midline abdominal incision. It was first described in 2001 by Rafi as a traditional blind landmark technique using the lumbar triangle of Petit. Local anesthetic is then injected between the internal oblique and transverse abdominis muscles just deep the fascial plane, the plane through which the sensory nerves pass

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 20-35 years
* Gestational age between 37-40 weeks
* Pregnant women undergoing elective cesarean section
* Medically free
* Singleton pregnancy

Exclusion Criteria:

* Emergency cesarean section
* Diabetic
* Hypertensive
* Severe anemia
* Multiple pregnancy
* Complication during section

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 400 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2022-03-20 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Post Operative Pain | 2 hours after the Cesarean Section till the pain relief
  The pain level of the cases is evaluated by means of the digital pain (numeric rating) scale from 0 to 10 in which 0 means "no pain" and 10 means "the worst pain" as well as the duration of pain relief

CONTACTS AND LOCATIONS:
Overall Officials: ElSayed ElDesouky, Professor, Principal Investigator — Al-Azhar University, Faculty of medicine for boys
Locations (1):
- Al-Azhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No